CLINICAL TRIAL: NCT00068107
Title: Study of Weekly Dosing Regimens of Replagal in Patients With Fabry Disease With Incomplete Clinical Response to Long-Term Therapy
Brief Title: Dosing Study of Replagal in Patients With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030286; 03-N-0286
Record Dates: First submitted 2003-09-06; First posted 2003-09-08 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Fabry Disease
Keywords: Lysosomal Storage; Renal Insufficiency; Stroke; Hypohidrosis; Peripheral Neuropathy; Fabry Disease
MeSH Terms: conditions — Fabry Disease; Renal Insufficiency; Stroke; Hypohidrosis; Peripheral Nervous System Diseases | interventions — agalsidase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Relagal (Experimental): All participants received Relagal administered weekly
  Interventions: Drug: Replagal

INTERVENTIONS:
Drug: Replagal — enzyme replacement therapy
  Other Names: agalsidase alfa

SUMMARY:
This study will determine the safety and effectiveness of increasing Replagal infusions in certain patients with Fabry disease. Replagal is a genetically engineered form of Alpha-galactosidase A, an enzyme that normally breaks down a fatty substance called globotriaosylceramide (Gb3). In patients with Fabry disease, Alpha-galactosidase A does not function properly and, therefore, Gb3 builds up, causing problems with the kidneys, heart, nerves, and blood vessels.

Patients with Fabry disease who are participating in NIH protocol 00-N-0185 or 02-N-0220 may be eligible for this study. This includes patients who are currently taking Replagal but whose kidney function continues to worsen, or patients who have certain test results that are much improved after Replagal infusion.

Participants will receive Replagal infusions (0.2 mg/kg body weight) through a vein once a week (as opposed to the previous dosage of once every 2 weeks) for up to 2 years. The first infusion, and some others, are given at the NIH Clinical Center, but most are administered by the patient's local doctor. Vital signs are measured before, immediately after, and 1 hour after each infusion.

Baseline evaluations are done on an inpatient basis at the NIH Clinical Center over a 1-week period before and after the first Replagal infusion and at 6-month intervals during the study. Tests include a check of vital signs (temperature, respiratory rate, pulse rate, and blood pressure); weight measurement; physical and neurological examinations; routine blood and urine tests; 24-hour urine collection; electrocardiogram; and review of treatment side effects. In addition, the following tests are done:

* Quantitative sensory testing: This is a non-invasive test to measure the ability to sense warm, cold and vibration in the hand and foot.
* QSART: This test measures the amount of sweat in a particular area of skin that did not sweat enough. A small amount of a medicine called acetylcholine is put on the skin and made to enter the skin using a very small electric current.
* Doppler skin blood flow: This test measures blood flow to the blood vessels of the skin. A machine takes pictures of blood flow in the skin of the forearm using a laser beam. Pictures are taken before and during application of medicines that cause blood vessels to dilate. Acetylcholine is used on one forearm and nitroprusside is used on the other. The medication is made to enter the skin using a small el...

DETAILED DESCRIPTION:
Objectives: The goal of this study is to determine whether higher frequency of dosing of enzyme replacement therapy (ERT) can either significantly slow the decline of renal function or continuously sustain the normalization of other objective functions in patients with Fabry disease who have been receiving intravenous infusions of Replagal (agalsidase alfa) at a dose of 0.2 mg/kg of body weight administered every 2 weeks.

Study Population: Patients with Fabry disease who are currently on clinical research protocols 00-N-0185/TKT011 or 02-N-0220/TKT015 and who have demonstrated progressive decline in calculated glomerular filtration rate (GFR) of at least 5 ml/min/year on ERT or who consistently show transient improvement in objective functions (such as sweating) in the few days post-infusion.

Design: This is an open label study comparing one dosing regimen with a previous less intensive dosing regimen. Patients will receive a dose of 0.2 mg/kg of body weight every week.

Outcome Measures: The main outcome measure will be a change in the mean linear rate of decline of the estimated calculated GFR. The main hypothesis is that a more frequent administration of the previous dose of Replagal will significantly reduce the mean slope of the decline of the calculated glomerular filtration rate GFR compared with the currently observed slope on a dose of 0.2 mg/kg administered every 2 weeks. At the 2-year time point, the dose will be increased to 0.4 mg/kg only in the patients whose GFR continues to significantly decline. Secondary outcome measures will be globotriaosylceramide (Gb(3)) in plasma and urinary sediment, quantitative sudomotor axon reflex test, quantitative sensory testing. Study duration is 2 years with a possibility of additional one-year extensions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with Fabry disease participating in 00-N-0185/TKT011 or 02-N-0220/TKT015 may be eligible. No other Fabry patients will be eligible.

Patients losing GFR at a rate greater than 5 ml/min/year despite ERT with agalsidase alfa for greater than or equal to 2.5 years in 00-N-0185/TKT/003/006/011 Study or ERT over greater than or equal to 1.0 years in 02-N-0220/TKT/010/015 Study.

Patients who at least twice demonstrated significant improvement or normalization of sweat function (by QSART or thermoregulatory sweat test) or reduction in serum creatinine by at least 10% but return to the pre-infusion state before the subsequent biweekly enzyme infusion.

Patients who freely agree to participate in this study and understand the nature, risks and benefits of this study and give their written informed consent.

EXCLUSION CRITERIA:

Patients with Fabry disease, who are not already part of 00-N-0185/TKT011 or 02-N-0220/TKT015.

Patients on these protocols who have stable serum creatinine (or a lesser rise in serum creatinine than stipulated in the inclusion criteria), and do not show other objective evidence of incomplete clinical response between biweekly infusions (e.g. sweat function).

Patients who have begun dialysis or who have received a renal transplant.

Patients who cannot tolerate the study procedures or who are unable or unwilling to travel to the study center as required by this protocol.

Patients with an intercurrent medical condition that would render them unsuitable for mthe study e.g. HIV, diabetes. The reason is that the pathologies of these conditions will be significant confounders in assessing the effect of the experimental therapy and its adverse events.

Patients who in the opinion of the investigator (for whatever reason) are thought to be unsuitable for the study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Altarescu G, Schiffmann R, Parker CC, Moore DF, Kreps C, Brady RO, Barton NW. Comparative efficacy of dose regimens in enzyme replacement therapy of type I Gaucher disease. Blood Cells Mol Dis. 2000 Aug;26(4):285-90. doi: 10.1006/bcmd.2000.0310. PMID 11042029
- [Background] Brady RO. Enzymatic abnormalities in diseases of sphingolipid metabolism. Clin Chem. 1967 Jul;13(7):565-77. No abstract available. PMID 5006481
- [Background] Brady RO, Schiffmann R. Clinical features of and recent advances in therapy for Fabry disease. JAMA. 2000 Dec 6;284(21):2771-5. doi: 10.1001/jama.284.21.2771. PMID 11105184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 participants were recruited; 1 participant was excluded because of stable kidney function; 12 started treatment
Groups:
- All Participants: All participants were followed on a prior protocol and found to have a mean slope on Replagal (agalsidase alfa) infused every 2 weeks of -0.66 +- 0.24 ml/min/month. Patients will receive a dose of 0.2 mg/kg of body weight every week.
Period: Overall Study
Arm/Group | All Participants
Started | 12
Completed | 3
Not Completed | 9
Not completed — end-stage renal disease | 6
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants were followed on a prior protocol and found to have a mean slope on Replagal (agalsidase alfa) infused every 2 weeks of -0.66 +- 0.24 ml/min/month.
Arm/Group | All Participants
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: The rate of decline in renal function, as measured by estimation of glomerular filtration rate at baseline when participants were receiving agalsidase alfa (Relagal) every 2 weeks and when participants were receiving weekly infusion of Relagal.
Time Frame: Relagal was administered every 2 weeks for 2-4 years pre-study, Relagal was administred weekly during the study (approx. 4.5-10 years)
Measure: Mean (Standard Deviation); unit: ml/min/month
Arm/Group | All Participants
Number analyzed (Participants) | 12
ml/min/month
  eGFR on infusions every 2 wks | -0.66 (0.24)
  eGFR on infusions weekly | -0.32 (0.34)
Statistical Analysis 1: Comparison: All Participants; eGFR measured pre-study was compared to eGFR during the study; Test type: Superiority or Other; p = 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: All Participants; Test type: Superiority or Other; Average Delay in time to ESRD = 166, 95% CI 2-sided [8.4 to 323.8] — The average delay in end stage renal disease (ESRD) calculated from the eGFR values and represents the estimated difference in time to ESRD between Relagal administered every 2 weeks and Relagal administered weekly. Units = months

2. Secondary Outcome: Globotriaosylceramide (Gb(3)) in Plasma
Time Frame: Baseline and last observation (up to 10 years)
Measure: Number; unit: nanomole/mL
Groups:
- All Participants at Baseline: All participants were followed on a prior protocol and found to have a mean slope on Replagal (agalsidase alfa) infused every 2 weeks of -0.66 +- 0.24 ml/min/month.
Arm/Group | All Participants at Baseline | All Participants at Last Observation
Number analyzed (Participants) | 11 | 11
nanomole/mL
  participant 1 | 2.35 | 4.10
  participant 2 | 4.62 | 5.58
  participant 3 | 2.43 | 2.62
  participant 5 | 3.17 | 3.60
  participant 6 | 6.78 | 5.04
  participant 7 | 3.32 | 3.21
  participant 8 | 3.69 | 4.51
  participant 9 | 4.25 | 1.91
  participant 10 | 2.59 | 3.41
  participant 11 | 6.62 | 5.62
  participant 12 | 6.56 | 6.63

3. Secondary Outcome: Globotriaosylceramide (Gb(3)) in Urine Sediment
Time Frame: Baseline and last observation (up to 10 years)
Measure: Number; unit: nanomole/(gram of Creatinine)
Arm/Group | All Participants at Baseline | All Participants at Last Observation
Number analyzed (Participants) | 11 | 11
nanomole/(gram of Creatinine)
  participant 1 | 49 | 1888
  participant 2 | 126 | 89
  participant 3 | 248 | 82
  participant 5 | 136 | 162
  participant 6 | 3026 | 652
  participant 7 | 3128 | 1682
  participant 8 | 1393 | 450
  participant 9 | 137 | 370
  participant 10 | 1457 | 488
  participant 11 | 2342 | 213
  participant 12 | 624 | 169

4. Secondary Outcome: Number of Participants With a Change in Quantitative Sudomotor Axon Reflex Test
Description: Quantitative sudomotor axon reflex test (QSART) is a measure of sweat function
Time Frame: Baseline and last observation (up to 10 years)
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 12
participants | 0

5. Secondary Outcome: Quantitative Sensory Testing
Description: For quantitative sensory testing, the outcome variable (detection threshold score) was analyzed for all combinations of location (foot, hand, and thigh) and test (cold, vibration, and warm). Possible threshold scores may range from 1-25. Score values of ">25" were set to 25. Higher scores indicate higher sensory detection threshold. Therefore, lower score is better. Time, measured in years, was centered at the date in which patients switched treatment regimen. All available measurements were used. A linear mixed model analysis was used to test for differences in the linear association between time and detection threshold score pre-and-post ERT regiment change while accounting for the correlation among observations from the same individual. Specifically, the model contained a subject specific random intercept with year as a fixed effect and knot at time of the treatment change.
Time Frame: pre-study was 2-4 years, during study sensory testing measured for approx. 4.5-5 years
Population: Number of participants with a sufficient number of data points to estimate slope
Measure: Mean (Standard Error); unit: units on a scale/year
Arm/Group | All Participants
Number analyzed (Participants) | 10
units on a scale/year
  Cold Sensory testing on Foot (pre-study) | -0.2108 (0.1366)
  Cold Sensory on Foot (difference pre- to post-) | 0.3863 (0.2784)
  Vibration Sensory testing on Foot (pre-study) | 0.3353 (0.1004)
  Vibration on Foot (difference pre- to post-) | -0.3912 (0.2041)
  Warm Sensory testing on Foot (pre-study) | -0.08536 (0.09264)
  Warm on Foot (difference pre- to post-) | 0.4169 (0.1887)
  Cold Sensory testing on Hand (pre-study) | -0.1026 (0.1413)
  Cold on Hand (difference pre- to post-) | 0.5141 (0.2874)
  Vibration Sensory testing on Hand (pre-study) | 0.2279 (0.07427)
  Vibration on Hand (difference pre- to post-) | -0.1966 (0.1503)
  Warm Sensory testing on Hand (pre-study) | -0.2138 (0.1179)
  Warm on Hand (difference pre- to post-) | 1.1781 (0.2401)
  Cold Sensory testing on Thigh (pre-study) | 0.2502 (0.1437)
  Cold on Thigh (difference pre- to post-) | -0.2991 (0.2884)
  Warm Sensory testing on Thigh (pre-study) | -0.549 (0.1124)
  Warm on Thigh (difference pre- to post-) | 0.8255 (0.2258)

6. Secondary Outcome: Doppler Skin Blood Flow
Time Frame: 10 years
Population: Doppler skin blood flow was not collected in this study because it was judged to not be useful early in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: All SAEs were adjudicated to be disease related and not related to the agalsidase alfa infusions.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 10/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=13)
catheter-induced peritonitis (Renal and urinary disorders) | 1
sepsis (Infections and infestations) | 1
hypotension (Cardiac disorders) | 1
advanced renal insufficiency (Renal and urinary disorders) | 1
myocardial infarction (Cardiac disorders) | 1
Sharp chest pain and right leg pain (Nervous system disorders) | 1
syncopal episode (Cardiac disorders) | 1 — occurred while straining when lifting weight in a gym
nausea and vomiting (General disorders) | 1
pain crisis (Nervous system disorders) | 1
elective mitral valve annuloplasty (Cardiac disorders) | 1
shortness of breath (Cardiac disorders) | 1
increased intensity of angina (Cardiac disorders) | 1
aortic stenosis (Cardiac disorders) | 1
ventricular tachycardia (Cardiac disorders) | 1
bacterial sepsis (Infections and infestations) | 1
recurrent ventricular arrhythmia (Cardiac disorders) | 1
hepatitis C infection (Infections and infestations) | 1
aortic valve replacement (Cardiac disorders) | 1
dizziness, tachycardia and chest pain (Cardiac disorders) | 1
severe renal decline (Renal and urinary disorders) | 1
clogged port-a-cath replacement and pacemaker adjustment (Cardiac disorders) | 1
placement of a pacemaker due to a bradycardic episode (Cardiac disorders) | 1
acute occipital ischemic stroke (Nervous system disorders) | 1
death (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=13)
Allergies (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 1
Arrythmia (Cardiac disorders) | 6
Impaired balance (General disorders) | 2
Blisters (Skin and subcutaneous tissue disorders) | 2
Burn (Skin and subcutaneous tissue disorders) | 1
Cancer - skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardiac palpitations (Cardiac disorders) | 1
Cholethisiasis (Gastrointestinal disorders) | 1
Cold symptoms (Infections and infestations) | 5
Creatinine worsened (Renal and urinary disorders) | 4
Depression (Psychiatric disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Dialysis (Renal and urinary disorders) | 3
Diaphoresis (General disorders) | 1
Dizziness (General disorders) | 1
Dreams (abnormal) (General disorders) | 1
Ecchymosis - varied (Skin and subcutaneous tissue disorders) | 1
Edema (Vascular disorders) | 2
Eosinophils - increased (Infections and infestations) | 1
Electrolytes - elevated (Renal and urinary disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 1
Ferritin - decreased (Blood and lymphatic system disorders) | 1
Ferritin - increased (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 2
Fracture (Musculoskeletal and connective tissue disorders) | 3
GI symptoms (Gastrointestinal disorders) | 2
Glucose - elevated (General disorders) | 1
Hair loss (General disorders) | 1
Headache (Nervous system disorders) | 2
Hearing Loss (Ear and labyrinth disorders) | 1
Heart Block (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Hypothyroid (Endocrine disorders) | 2
Infection (Infections and infestations) | 3
Injury - trauma (Injury, poisoning and procedural complications) | 1
Iron - decreased (Blood and lymphatic system disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Kidney nodules/cysts (Renal and urinary disorders) | 1
Malaise (General disorders) | 1
Memory - decreased (Nervous system disorders) | 1
Mental status altered (Nervous system disorders) | 1
Microalbuminuria - worsened (Renal and urinary disorders) | 3
Numbness (Nervous system disorders) | 1
Orthopedic (Musculoskeletal and connective tissue disorders) | 1
Pain - back (General disorders) | 1
Pain - chest (no specific angina) (General disorders) | 3
Pain - finger (General disorders) | 1
Pain - GI (General disorders) | 2
Pain - knee (General disorders) | 2
Pain - leg (spastic) (General disorders) | 1
Pain - neck area (General disorders) | 2
Pain - pelvic area (General disorders) | 1
Pain - shoulder (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Potassium - elevated (Blood and lymphatic system disorders) | 3
Proteinuria - increased (Renal and urinary disorders) | 4
Prostatic hypertrophy (Renal and urinary disorders) | 1
Prostatitis (Renal and urinary disorders) | 1
PSA - elevated (General disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Renal failure (Renal and urinary disorders) | 3
Restless Leg Syndrome (Nervous system disorders) | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Infection (Infections and infestations) | 2
Sodium - elevated (Blood and lymphatic system disorders) | 1
Speech - impaired (Nervous system disorders) | 1
Stool leakage (Gastrointestinal disorders) | 1
Stroke - acute ischemic (Nervous system disorders) | 1
Throat - dry (General disorders) | 1
Transplant - kidney (Renal and urinary disorders) | 1
Tremors (Nervous system disorders) | 1
TSH - elevated (Endocrine disorders) | 1
Urine - bloody s/p prostate biopsy (Renal and urinary disorders) | 1
Virus - post transplant (General disorders) | 1
Vision - hazy (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight loss - unexpected (General disorders) | 2

LIMITATIONS AND CAVEATS:
Small number of subjects. Single group with comparison to baseline data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No